CLINICAL TRIAL: NCT04177823
Title: A Phase I Open-label, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Clinical Activity of the Antibody Drug Conjugate GSK2857916 in Chinese Participants With Relapsed/Refractory Multiple Myeloma Who Have Failed At Least Two Lines of Previous Treatment, Containing an Alkylator, a Proteasome Inhibitor and an Immunomodulatory Agent
Brief Title: A Study of Belantamab Mafodotin to Investigate Safety, Tolerability, Pharmacokinetics, Immunogenicity and Clinical Activity in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208465
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: belantamab mafodotin; DLT; RRMM
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Intervention Model Description: This study has 3+3 dose escalation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chinese participants with relapsed/refractory multiple myeloma (Experimental): Participants will be administered belantamab mafodotin 2.5 mg/kg or 3.4 mg/kg as an intravenous infusion on Day 1 of each 21-day cycle over 30 minutes. Participants will be treated until disease progression, intolerable toxicity, end of study or informed consent withdrawal.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be available as lyophilized powder 100 mg/vial in single-use vial for reconstitution. It will be administered at a calculated dose of 2.5 mg/kg or 3.4 mg/kg as an IV infusion on Day 1 of each cycle over 30 minutes.

SUMMARY:
Multiple myeloma (MM) is a neoplastic plasma cell disorder that is characterized by osteolytic bone lesions, anemia, hypercalcemia and renal failure. belantamab mafodotin was well tolerated in previous studies with at least one dose of belantamab mafodotin in heavily pre-treated participants with relapsed/refractory multiple myeloma (RRMM). This aim of the study is to explore safety, pharmacokinetics (PK), tolerability, immunogenicity and clinical activity of belantamab mafodotin monotherapy in Chinese participants with RRMM who have received at least 2 prior line of anti-myeloma therapy including an alkylator, a proteasome inhibitor (PI) and an immunomodulatory agent (IMiD). This study will include two dose cohorts 2.5 milligram per kilogram (mg/kg) and 3.4 mg/kg. A maximum of 12 participants will be enrolled, 6 each for 2.5 mg/kg cohort and 3.4 mg/kg cohort based on 3+3 design. Participants will be treated until disease progression, intolerable toxicity, end of study or informed consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent, which includes compliance with requirements and restrictions listed in the consent form.
* Male or female, 18 years or older (at the time consent is obtained).
* Eastern Cooper Oncology Group (ECOG) performance status of 0-2.
* Histological or cytologically confirmed diagnosis of MM as defined according to IMWG criteria and a) Has undergone stem cell transplant or transplant is considered not feasible by local assessment, b) Has failed at least 2 prior lines of anti-myeloma treatments, containing all of the following classes of drugs: alkylating agent, IMID and PI, c) In addition, eligible participant needs to be refractory to an IMiD (i.e.,lenalidomide or pomalidomide), and to a proteasome inhibitor (i.e., bortezomib, ixazomib or carfizomib) as defined by International Myeloma Working Group (IMWG) criteria, d) Participants who failed with cluster of differentiation38 (CD38) antibody (i.e., daratumumab) in previous clinical trials can also be considered to include if they meet the remainder of inclusion criteria in this protocol.
* Has measurable disease with at least one of the following: a) Serum M-protein greater than or equal to 0.5 grams per deciliter (g/dL) (5 g/L) , b) Urine M-protein greater than or equal to 200 mg/24hour, c) Serum Free light chain (FLC) assay: Involved FLC level greater than or equal to10 mg/dL (greater than or equal to 100 mg/L) and an abnormal serum free light chain ratio (less than 0.26 or greater than 1.65)
* Participants with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met: a) Transplant was greater than 100 days prior to study enrolment, b) No active infection(s), c) Participant meets the remainder of the eligibility criteria outlined in this protocol.
* Adequate organ system functions.
* Female Participants: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of less than 1 percent per year), preferably with low user dependency, during the intervention period and for at least 80 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Male Participants: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 140 days: Refrain from donating sperm, plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. or Must agree to use contraception/barrier as detailed below: Agree to use a male condom and female partner to use an additional highly effective contraceptive method with a failure rate of less than 1 percent per year as when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* All prior treatment-related toxicities (defined by National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0 must be less than or equal to Grade 1 at the time of enrolment except for alopecia and Grade 2 peripheral neuropathy.

Exclusion Criteria:

* Systemic anti-myeloma therapy within less than 14 days, or plasmapheresis within 7 days prior to the first dose of study drug.
* Symptomatic amyloidosis, active polyneuropathy,organomegaly, endocrinopathy, myeloma protein, and skin changes (POEMS) syndrome, active plasma cell leukemia at the time of screening.
* Prior allogeneic stem cell transplant (SCT).
* Current corneal epithelial disease except mild punctate keratopathy.
* Use of an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs. Prior B-cell maturation antigen (BCMA) targeted therapy.
* Evidence of active mucosal or internal bleeding.
* Any major surgery within the last four weeks.
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil criteria.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Malignancies other than disease under study are excluded, except for any other malignancy from which the participant has been disease-free for more than 2 years and, in the opinion of the principal investigators and GSK Medical Monitor, will not affect the evaluation of the effects of this clinical trial treatment on the currently targeted malignancy (MM).
* Evidence of cardiovascular risk including any of the following: a) corrected QT internal Fridericia (QTcF) interval greater than equal to 480 milliseconds (msecs), b) Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block, c) History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three months of Screening, d) Class III or IV heart failure as defined by the New York Heart Association functional classification system, e) Uncontrolled severe hypertension, e.g. 170/110.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin, or any of the components of the study intervention.
* Pregnant or lactating female.
* Active infection requiring antibiotic, antiviral, or antifungal treatment.
* Known human immunodeficiency virus (HIV) infection.
* Presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb at screening or within 3 months prior to first dose of study intervention).
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beijing, China

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not randomized to 3.4 mg/kg dose or de-escalated to the 1.9 mg/kg dose
Groups:
- Belantamab Mafodotin: Participants with relapsed/refractory multiple myeloma (RRMM) were administered with 2.5 milligram per kilogram (mg/kg) belantamab mafodotin intravenous (IV) infusion over 30-60 minutes on day 1 of each 21-days cycle. Participants were treated until disease progression, intolerable toxicity, end of study or informed consent withdrawal.
Period: Overall Study
Arm/Group | Belantamab Mafodotin
Started | 6
Completed | 4
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 24 months and 21 days
Population: All treated population included all eligible participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; important medical events that may jeopardize the participant or may require medical or surgical intervention; is associated with liver injury and impaired liver function.
Time Frame: Up to 24 months and 21 days
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants | 1

3. Primary Outcome: Number of Participants With Dose Limited Toxicities (DLTs)
Description: An event was considered DLT if it occurred within 21 days of treatment and met any of the following criteria within same period:
  * Any Grade (Gr.) 3 or greater non-hematologic toxicity as described in NCI-CTCAE Version 5.0, other than corneal events that persists for >48 hours despite supportive treatment or leads to hospitalization.
  * Hematologic toxicity such as Gr. 3 or greater febrile neutropenia lasting >48 hours despite adequate treatment (Gr. 3 defined as absolute neutrophil count (ANC) <1000/millimeter cube (mm^3) at a single temperature >38.3 degree celsius or a sustained temperature >=38 degree celsius for more than 1 hour) and, Gr. 4 thrombocytopenia defined as platelet count <25000/mm^3 with clinically significant bleeding, or if platelet transfusion is required.
  * Gr. 4 per the corneal grading scale.
  * Liver toxicity meeting pre-specified by GSK liver stopping criteria.
Time Frame: Day 1 to day 21 of cycle 1
Population: DLT evaluable population included all the eligible participants who have received the 1st dose as planned and experienced a DLT during the cycle 1 or completed the cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC[0-t]) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of belantamab mafodotin. PK parameters were analyzed using standard non-compartmental analysis. AUC[0-t] was calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: Pre-dose (within 30 minutes prior to start of infusion), end of infusion (EOI), 2, 4, 8 and 24 hours post start of infusion (HPS) on day 1, anytime on day 2, 4, 8, 15 and 22 of cycle 1 (each cycle is of 21 days)
Population: Pharmacokinetic (PK) population, was defined as those participants in the "All treated" population from whom at least one PK sample was obtained, analyzed, and was measurable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter (h*ug/mL)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hours*microgram per milliliter (h*ug/mL) | 2819.39 (30.32)

5. Secondary Outcome: AUC[0-t] of Belantamab Mafodotin Total Antibody
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
h*ug/mL | 5407.64 (33.03)

6. Secondary Outcome: AUC[0-t] of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hours*nanograms per milliliter (h*ng/mL) | 136.17 (48.66)

7. Secondary Outcome: Area Under the Concentration-time Curve During the Dosing Interval (AUC[0-tau]) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of belantamab mafodotin. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
h*ug/mL | 2853.73 (28.81)

8. Secondary Outcome: AUC[0-tau] of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
h*ug/mL | 4823.61 (20.56)

9. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 168h (AUC[0-168]) of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 7
Time Frame: Up to 168 hours
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
h*ng/mL | 133.94 (53.14)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0-infinity]) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
h*ug/mL | 3000.34 (35.32)

11. Secondary Outcome: AUC[0-infinity] of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
h*ug/mL | 5514.32 (29.69)

12. Secondary Outcome: AUC[0-infinity] of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 3
h*ng/mL | 172.75 (62.22)

13. Secondary Outcome: Observed Plasma Concentration at the End of Infusion (CEOI) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: Pre-dose (within 30 minutes prior to start of infusion) on day 1 of cycle 2, 4, 6, 9 and 12 (each cycle is of 21 days)
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (ug/mL)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Micrograms per milliliter (ug/mL)
  Cycle 1 | 41.50 (59.71)
  Cycle 2: number analyzed (Participants) | 5
  Cycle 2 | 36.99 (76.89)
  Cycle 4: number analyzed (Participants) | 3
  Cycle 4 | 41.76 (17.35)
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 43.69 (7.61)
  Cycle 9: number analyzed (Participants) | 1
  Cycle 9 | 40.10
  Cycle 12: number analyzed (Participants) | 1
  Cycle 12 | 33.20

14. Secondary Outcome: CEOI of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: Pre-dose (within 30 minutes prior to start of infusion) on day 1 of cycle 2, 4, 6, 9 and 12 (each cycle is of 21 days)
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
ug/mL
  Cycle 1 | 33.78 (48.20)
  Cycle 2: number analyzed (Participants) | 4
  Cycle 2 | 60.36 (47.69)
  Cycle 4: number analyzed (Participants) | 3
  Cycle 4 | 58.75 (26.32)
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 67.70 (1.67)
  Cycle 9: number analyzed (Participants) | 1
  Cycle 9 | 66.00
  Cycle 12: number analyzed (Participants) | 1
  Cycle 12 | 64.70

15. Secondary Outcome: CEOI of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 7
Time Frame: Pre-dose (within 30 minutes prior to start of infusion) on day 1 of cycle 2, 4, 6, 9 and 12 (each cycle is of 21 days)
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Nanograms per milliliter (ng/mL)
  Cycle 1 | 0.53 (80.68)
  Cycle 2: number analyzed (Participants) | 5
  Cycle 2 | 0.74 (75.24)
  Cycle 4: number analyzed (Participants) | 3
  Cycle 4 | 0.44 (19.63)
  Cycle 6: number analyzed (Participants) | 2
  Cycle 6 | 0.47 (10.34)
  Cycle 9: number analyzed (Participants) | 1
  Cycle 9 | 0.37
  Cycle 12: number analyzed (Participants) | 1
  Cycle 12 | 0.38

16. Secondary Outcome: Maximum Observed Concentration (Cmax) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of belantamab mafodotin. PK parameters were analyzed using standard non-compartmental analysis. Maximum observed plasma concentration, determined directly from the concentration-time data for each cycle.
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
ug/mL | 45.36 (54.69)

17. Secondary Outcome: Cmax of Belantamab Mafodotin Total Antibody
Description: as for outcome 16
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
ug/mL | 42.21 (19.65)

18. Secondary Outcome: Cmax of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 16
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
ng/mL | 1.41 (51.14)

19. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hour | 2.03 [0.6 to 2.2]

20. Secondary Outcome: Tmax of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hour | 2.03 [1.0 to 2.2]

21. Secondary Outcome: Tmax of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hour | 7.96 [0.6 to 46.6]

22. Secondary Outcome: Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hour | 504.54 [329.8 to 509.9]

23. Secondary Outcome: Tlast of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hour | 507.23 [478.2 to 545.7]

24. Secondary Outcome: Tlast of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Hour | 168.15 [162.0 to 336.0]

25. Secondary Outcome: Systemic Clearance (CL) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
Liter per hour (L/h) | 0.0518 (27.29)

26. Secondary Outcome: CL of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
L/h | 0.0300 (25.15)

27. Secondary Outcome: Systemic Clearance Normalized by Body Weight (CL/Weight) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour per kilogram
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
Milliliter per hour per kilogram | 0.83 (35.94)

28. Secondary Outcome: CL/Weight of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour per kilogram
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
Milliliter per hour per kilogram | 0.46 (29.08)

29. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
Liter (L) | 7.57 (10.63)

30. Secondary Outcome: Vss of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
L | 6.62 (19.63)

31. Secondary Outcome: Volume of Distribution at Steady State Normalized by Body Weight (Vss/Weight) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per kilogram (mL/kg)
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
Milliliter per kilogram (mL/kg) | 122.11 (18.60)

32. Secondary Outcome: Vss/Weight of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
mL/kg | 101.41 (15.58)

33. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 5
Hour | 128.25 (23.52)

34. Secondary Outcome: t1/2 of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 4
Hour | 169.20 (18.34)

35. Secondary Outcome: t1/2 of Belantamab Mafodotin Cys- Monomethyl Auristatin-F (Cys-mcMMAF)
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 3
Hour | 73.61 (18.33)

36. Secondary Outcome: Trough Concentration Prior to the Next Dose for Each Cycle (Ctrough) of Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: as for outcome 7
Time Frame: Pre-dose (within 30 minutes prior to start of infusion) on day 1 of cycle 1, 3, 5, 8 and 11 (each cycle is of 21 days)
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
ug/mL
  Cycle 1: number analyzed (Participants) | 5
  Cycle 1 | 1.14 (73.76)
  Cycle 3: number analyzed (Participants) | 3
  Cycle 3 | 2.43 (104.26)
  Cycle 5: number analyzed (Participants) | 2
  Cycle 5 | 5.70 (4.09)
  Cycle 8: number analyzed (Participants) | 1
  Cycle 8 | 4.59
  Cycle 11: number analyzed (Participants) | 1
  Cycle 11 | 4.41

37. Secondary Outcome: Ctrough of Belantamab Mafodotin Total Antibody
Description: as for outcome 7
Time Frame: Pre-dose (within 30 minutes prior to start of infusion) on day 1 of cycle 1, 3, 5, 8 and 11 (each cycle is of 21 days)
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
ug/mL
  Cycle 1: number analyzed (Participants) | 5
  Cycle 1 | 3.76 (79.96)
  Cycle 3: number analyzed (Participants) | 3
  Cycle 3 | 10.25 (105.86)
  Cycle 5: number analyzed (Participants) | 2
  Cycle 5 | 24.50 (1.15)
  Cycle 8: number analyzed (Participants) | 1
  Cycle 8 | 23.90
  Cycle 11: number analyzed (Participants) | 1
  Cycle 11 | 26.40

38. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Abnormal vital signs were defined as any abnormal findings in the vital signs parameters (temperature, blood pressure and pulse rate).
Time Frame: Up to 21 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants | 0

39. Secondary Outcome: Number of Participants With Worst- Case Grade Changes Post-baseline in Hematology Parameter: Hemoglobin, Lymphocytes, Neutrophils, Platelets, Leukocytes
Description: Blood samples were collected at indicated time points to assess change from baseline in hemoglobin, lymphocytes, neutrophils, platelets, leukocytes. Worst case grade increase from baseline grade was provided for all the hematology tests that were gradable by National Cancer Institute Common Terminology Criteria (NCI CTCAE, Version 5.0, 2017). Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE. Data for any participants with worst-case grade changes (Increase to Grade 3 or Increase to Grade 4) post-baseline were presented. Baseline was defined as latest pre-dose assessment (day 1) with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (day 1) and up to 21 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants
  Hemoglobin, increase to grade 3 | 2
  Hemoglobin, increase to grade 4 | 0
  Lymphocytes, increase to grade 3 | 0
  Lymphocytes, increase to grade 4 | 0
  Neutrophils, increase to grade 3 | 1
  Neutrophils, increase to grade 4 | 0
  Platelets, increase to grade 3 | 1
  Platelets, increase to grade 4 | 1
  Leukocytes, increase to grade 3 | 1
  Leukocytes, increase to grade 4 | 0

40. Secondary Outcome: Number of Participants With Worst- Case Grade Changes Post-baseline in Clinical Chemistry Parameters
Description: Blood samples were collected at indicated time points to assess change from baseline in albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, bilirubin, creatine kinase, gamma glutamyl transferase, potassium, lactate dehydrogenase, magnesium. Worst case grade (G) increase from baseline grade was provided for all the chemistry tests that were gradable by National Cancer Institute Common Terminology Criteria (NCI CTCAE, Version 5.0, 2017). Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE. Data for any participants with worst-case grade changes (Increase to Grade 3 or Increase to Grade 4) post-baseline were presented. Baseline was defined as latest pre-dose assessment (day 1) with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (day 1) and up to 21 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants
  Albumin, increase to G3 | 0
  Albumin, increase to G4 | 0
  Alkaline Phosphatase, increase to G3 | 0
  Alkaline Phosphatase, increase to G4 | 0
  Alanine Aminotransferase, increase to G3 | 0
  Alanine Aminotransferase, increase to G4 | 0
  Aspartate Aminotransferase, increase to G3 | 0
  Aspartate Aminotransferase, increase to G4 | 0
  Bilirubin, increase to G3 | 0
  Bilirubin, increase to G4 | 0
  Creatine Kinase, increase to G3 | 0
  Creatine Kinase, increase to G4 | 0
  Gamma Glutamyl Transferase, increase to G3 | 0
  Gamma Glutamyl Transferase, increase to G4 | 0
  Potassium, increase to G3 | 0
  Potassium, increase to G4 | 0
  Lactate Dehydrogenase, increase to G3 | 0
  Lactate Dehydrogenase, increase to G4 | 0
  Magnesium, increase to G3 | 0
  Magnesium, increase to G4 | 0

41. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed partial response (PR) or better (i.e., very good partial response [VGPR], complete response [CR] and stringent complete response [sCR]) as assessed by International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma 2016. PR=response greater than or equal to (>=) 50 percent (%) reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to less than (<) 200 mg per 24 hours. CR=negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. sCR=complete response below plus normal free light chain (FLC) ratio and absence of clonal plasma cells in bone marrow by immunohistochemistry or 8-color, 2 tube multiparametric flow cytometry. VGPR=Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-component level <100 mg/24 h.
Time Frame: Up to 21 months
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Percentage of Participants | 16.7 [0.4 to 64.1]

42. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples were analyzed for the presence of anti-belantamab mafodotin antibodies by a validated electro chemiluminescent immunoassay. All samples were tested in a screening assay to identify potentially positive samples.
Time Frame: Up to 24 months and 21 days
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Participants | 1

43. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Samples were analyzed for the presence of anti-belantamab mafodotin antibodies by a validated electro chemiluminescent immunoassay. All samples were tested in a screening assay to identify potentially positive samples. Screened positive was further characterized for the antibody titer values.
Time Frame: Up to 24 months and 21 days
Population: All Treated Population. Only the participants who showed positive results for ADAs were analyzed.
Measure: Number; unit: Titer
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 1
Titer | 100

44. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total Score
Description: The OSDI instrument measures vision-related function. The total OSDI score was calculated as (sum of scores for all questions answered*100) divided by (total number of questions answered*4). The 12 items questionnaire assessed ocular symptoms, visual-related functioning and environmental triggers. Scores ranged from 0 to 100, with higher scores indicating a worse status. Baseline was defined as latest pre-dose assessment (day 1) with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (day 1) Up to 24 months and 21 days
Population: All treated population
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Belantamab Mafodotin
Number analyzed (Participants) | 6
Scores on Scale | 12.8 (20.43)

ADVERSE EVENTS:
Time Frame: All cause mortality, Non-serious adverse events (Non-SAEs) and serious adverse events (SAE) were collected for up to 24 months and 21 days
Description: All treated population included all eligible participants who received at least 1 dose of study treatment.
Arm/Group | Belantamab Mafodotin
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin (N=6)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin (N=6)
Platelet count decreased (Investigations) | 4 (10)
Blood lactate dehydrogenase increased (Investigations) | 4 (7)
Lymphocyte count decreased (Investigations) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Neutrophil count decreased (Investigations) | 3 (5)
White blood cell count decreased (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 2 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (3)
Adenosine deaminase increased (Investigations) | 1 (2)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (2)
Glycocholic acid increased (Investigations) | 1 (2)
Protein total decreased (Investigations) | 1 (2)
Crystal urine present (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Leucine aminopeptidase increased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Prealbumin decreased (Investigations) | 1 (1)
Total bile acids increased (Investigations) | 1 (1)
Urinary occult blood (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Punctate keratitis (Eye disorders) | 2 (3)
Vision blurred (Eye disorders) | 2 (3)
Visual impairment (Eye disorders) | 1 (1)
Pyrexia (General disorders) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04177823/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04177823/SAP_001.pdf